CLINICAL TRIAL: NCT03900286
Title: Evaluating the Therapeutic Efficacy and Metabolic Impact of a Low Energy Diet (LED) in People With Familial Partial Lipodystrophy and Diabetes
Brief Title: Low Energy Diet and Familial Partial Lipodystrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mandour Omer Mandour, Wellcome Trust Senior Clinical Fellow, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A095183
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Lipodystrophy; Diabetes; Diet Modification
Keywords: Familial Partial Lipodystrophy; FPLD; Diet; Total Diet Replacement; Diabetes
MeSH Terms: conditions — Lipodystrophy; Diabetes Mellitus; Lipodystrophy, Familial Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): Total Diet Replacement for 12 weeks, food reintroduction 6 weeks
  Interventions: Dietary Supplement: Total Dietary Replacement

INTERVENTIONS:
Dietary Supplement: Total Dietary Replacement — Total Dietary Replacement

SUMMARY:
To evaluate the therapeutic efficacy and metabolic impact of a low energy diet (LED) in people with familial partial lipodystrophy and diabetes. Participants will be provided with a LED (total diet replacement) for 12 weeks, before the introduction of a stepped food transition. Metabolic effects will continue to be assessed for 1 year. In order to better understand why this intervention changes insulin sensitivity, we will also collect adipose and muscle tissue samples at baseline and 12 weeks into the intervention in participants willing to have these procedures performed. These samples will be used for histological, metabolite, gene expression and protein expression analyses.

ELIGIBILITY:
Inclusion Criteria:

* Familial Partial Lipodystrophy
* Age >= 18 yrs
* T2DM
* Willingness to check daily blood sugars
* HbA1c between 53mmol(7%)- 108 mmol(12%)
* Weight stable for 3 months
* Capacity to consent

Exclusion Criteria:

* Pregnancy
* Untreated thyroid dysfunction (patients who have been euthyroid on medication for at least 3 months can be included)
* Use of medication adversely that affects diabetes control (e.g. steroids/ immunosuppressants/ certain antipsychotics)
* Incapacity to give informed consent
* History of an eating disorder/ purging behaviour
* Previous gastric bypass/ banding
* Use of Leptin Therapy
* Untreated retinopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
A change from baseline in HbA1c | 12 weeks
  mmol/mol

SECONDARY OUTCOMES:
A change from baseline in HbA1c | 1 year
  mmol/mol
A change from baseline in fasting glucose | 12 weeks, 1 year
  mmol/l
A change from baseline in triglycerides | 12 weeks, 1 year
  mmol/l
A change from baseline in liver fat | 12 weeks, 1 year
  % liver fat on MRI
A change from baseline in pancreatic fat | 12 weeks, 1 year
  % pancreatic fat on MRI
A change from baseline in insulin sensitivity | 12 weeks, 1 year
  Insulin pmol/l values during oral glucose tolerance test
A change from baseline in quality of life scores | 12 weeks, 1 year
  Change in scores of EQ-5D-3L Quality of Life measurement from baseline. EQ-5D-3L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life.
  It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
  This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
A change from baseline in anxiety scores | 12 weeks, 1 year
  Change in scores of Generalised Anxiety Disorder-7 (GAD 7) from baseline. Change in scores of Generalised Anxiety Disorder-7 (GAD 7) from baseline. The Generalised Anxiety Disorder-7 (GAD 7) Questionnaire is a 7 item measurement that is used to measure or assess the severity of generalised anxiety disorder (GAD)
  The index scores are as follows:
  0 - 4 No Anxiety 5 - 10 Mild Anxiety 11 - 15 Moderate Anxiety 15 - 21 Severe Anxiety
A change from baseline in depression scores | 12 weeks, 1 year
  Change in scores of Patient Health Questionnaire-9 (PHQ9), from baseline. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  The responses for each of the 9 items are:
  * 0 - Not at all
  * 1 - Several days
  * 2 - More than half the day
  * 3 - Nearly every day
  The score ranges are:
  0 - 4 None 5 - 9 Mild 10 - 14 Moderate 15 - 19 Moderately Severe 20 - 27 Severe
A change from baseline in antidiabetic medication use | 12 weeks, 1 year
  A change in the amount of antidiabetic drugs taken and/or a change in dose.
Adult Eating Behaviour Questionnaire | 12 weeks, 1 year
  Change in scores in eating behaviour
The Three Factor Eating Questionnaire | 12 weeks, 1 year
  Change in scores in The Three Factor Eating Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Savage, Principal Investigator — Wellcome Trust-MRC Institute of Metabolic Science, University of Cambridge
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim EL, Hollingsworth KG, Aribisala BS, Chen MJ, Mathers JC, Taylor R. Reversal of type 2 diabetes: normalisation of beta cell function in association with decreased pancreas and liver triacylglycerol. Diabetologia. 2011 Oct;54(10):2506-14. doi: 10.1007/s00125-011-2204-7. Epub 2011 Jun 9. PMID 21656330
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645

DOCUMENTS (1):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03900286/Prot_000.pdf